CLINICAL TRIAL: NCT04715165
Title: Comparison of Subcostal Transversus Abdominis Block With Intraperitoneal Instillation of Bupivacaine and Dexmedetomidine for Pain Relief After Laparoscopic Cholecystectomy: A Randomized Trial
Brief Title: Analgesia After Laparoscopic Cholecystectomy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Seham Mohamed Moeen Ibrahim, Assiut University, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SM 1, 2021
Record Dates: First submitted 2021-01-15; First posted 2021-01-20 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-08

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Active Comparator): Patients will receive USG-STAP block with bupivacaine and dexmedetomidine in both sides ten minutes before skin incision and intraperitoneal normal saline.
  Interventions: Drug: USG-STAP with bupivacaine and dexmedetomidine
- Group II (Placebo Comparator): Patients will receive bupivacaine and dexmedetomidine through the intraperitoneal route and USG-STAP block with normal saline at the end of surgery
  Interventions: Drug: IP bupivacaine and dexmedetomidine

INTERVENTIONS:
Drug: USG-STAP with bupivacaine and dexmedetomidine — Patients will receive USG-STAP block with bupivacaine and dexmedetomidine in both sides ten minutes before skin incision and intraperitoneal normal saline
  Arms: Group I
Drug: IP bupivacaine and dexmedetomidine — Patients will receive bupivacaine and dexmedetomidine through the intraperitoneal route and USG-STAP block with normal saline at the end of surgery
  Arms: Group II

SUMMARY:
Pain after laparoscopic cholecystectomy is common and may lead to delayed hospital discharge.

DETAILED DESCRIPTION:
Laparoscopic cholecystectomy (LC) is very commonly performed nowadays, and it has now completely replaced open cholecystectomy in the management of biliary lithiasis. Although it is minimally invasive surgery, pain in postoperative period is always major concern as it increases perioperative stress, morbidity, and hospital stay.

There are two components involved in pain after LC; the visceral component is due to tissue damage in anterior abdominal wall during the insertion of trocar and shoulder tip pain due to diaphragmatic irritation caused by Spillage of blood or bile and peritoneum stretching caused by pneumoperitoneum.

There are several methods employed in the management of postoperative pain after LC such as conventional systemic analgesics, including paracetamol, non-steroidal anti-inflammatory drugs, systemic opioids, thoracic epidural analgesia, low-pressure pneumoperitoneum, and warm air with all having its side effects .

Transversus abdominis plane (TAP) block has got a substantial role in postoperative analgesia after abdominal surgery because deposition of local anesthetics in transversus abdominis fascial plane can produce sensory block over the anterior abdominal wall from T7 to L1. Many clinical studies reported beneficial effects of TAP but results were mainly connected to lower abdominal surgery. Since the major part of pain after LC derives from abdominal wall incisions, some trials investigated TAP block as potential analgesic option. Some studies showed that TAP block can reduce opioid requirements and pain scores but the results were not conclusive enough because many differences in study designs.

The ultrasound-guided (USG) subcostal transversus abdominis plane block (STAP), first described by Hebbard 2008, is a variation of TAP which successfully solve the problem of unreliable supraumbilical distribution of the block. Results obtained in a few small studies showed significantly better analgesia after LC compare to traditional opioid analgesia, port-site infiltration and standard TAP.

Intraperitoneal (IP) instillation of local anaesthetics around the operative site is used as an analgesic technique on the assumption that conduction from visceral sites is obstructed and may lessen the intensity of referred pain to the shoulder (C3, C4) which results from irritation of diaphragmatic innervations, i.e., phrenic nerve (C3, C4, C5) and diaphragmatic stretching due to gaseous distension, in the postoperative period. Narchi I' et al., as early as in 1991 had reported that instillation of local anaesthetic (80 mL of bupivacaine 0.125%, epinephrine (1:200,000) under the right diaphragm reduced shoulder pain after minor gynaecologic laparoscopy.

Dexmedetomidine is a selective, short acting, agonist of the α2-adrenergic receptors. It has high affinity to α2-adrenergic receptors (more than eight-fold) and lower affinity to α1-receptors, compared with other α2-agonists agents, besides its great selectivity to α2A-adrenergic receptors, which is responsible for its analgesic effect. It has been used clinically as an adjunct to anesthesia and analgesia, and it is useful for painful surgical procedure and ICU sedation.

ELIGIBILITY:
Inclusion Criteria:

• Patients undergoing elective LC under general anesthesia, aged from 20 to 65 years old.

Exclusion Criteria:

* Contraindications to regional block (coagulopathy, infection at the needle insertion site, or diaphragmatic paralysis)
* Altered conscious level
* Pregnancy
* Body mass index (BMI > 35)
* Patients who have difficulty understanding the study protocol 6- Patients who have any known contraindication to study medications 7- Patient refusal.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-08-07 (Actual); Primary Completion 2022-02-15 (Estimated); Study Completion 2022-02-15 (Estimated)

PRIMARY OUTCOMES:
The intensity of postoperative pain | 24 hours after surgery
  Assessed by the numerical rating pain scale (NRS)

CONTACTS AND LOCATIONS:
Overall Officials: Seham M Moeen, MD, Principal Investigator — Assiut University
Locations (1):
- Assiut University, Asyut, Egypt

REFERENCES:
- [Derived] El Sabour AIA, Youssef HA, Ismail EA, Ahmed DH. Comparison of subcostal transversus abdominis block with intraperitoneal instillation of bupivacaine and dexmedetomidine for pain relief after laparoscopic cholecystectomy, randomized double blinded controlled study. BMC Anesthesiol. 2025 Nov 14;25(1):560. doi: 10.1186/s12871-025-03412-4. PMID 41239226